CLINICAL TRIAL: NCT06193980
Title: Exercise Testing in ICU Survivors to Evaluate ICU-acquired Weakness
Brief Title: ICU Combined Assessment of Cardio-Respiratory Exercise
Acronym: ICU-CARE
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Asher Mendelson, Assistant Professor, University of Manitoba
Other Study IDs: HS25592
Record Dates: First submitted 2023-12-08; First posted 2024-01-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: ICU Acquired Weakness; Sepsis; Shock; Critical Illness; Microcirculation
Keywords: ICU Survivors; Oxygen Delivery; Microcirculation; skeletal muscle; Exercise; near-infrared spectroscopy; cardiopulmonary exercise test; cardiovascular physiology
MeSH Terms: conditions — Sepsis; Shock; Critical Illness; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU survivors: Patients who have received prolonged mechanical ventilation (7 days or more) in the intensive care unit (ICU), and have been discharged from hospital.

SUMMARY:
This study aims to investigate how sepsis and critical illness can impair the cardiovascular system and microcirculation in intensive care unit (ICU) patients, which can lead to long-lasting muscle weakness/dysfunction or ICU-Acquired Weakness (ICU-AW) and exercise limitations.

DETAILED DESCRIPTION:
This longitudinal study will assess cardiovascular fitness and microvascular function through two (2) follow-ups after ICU discharge: at (i) 6 months, and (ii) 12 months. The goal is to understand how microvascular dysfunction contributes to ICU-AW and long-term exercise limitation in ICU survivors.

Specific goals are:

1. Evaluate peak oxygen uptake and oxygen on/off kinetics in ICU survivors using a standardized cardiopulmonary exercise test (CPET) protocol.
2. Characterize skeletal muscle microvascular function in ICU survivors using high-resolution NIRS during CPET protocol.
3. Determine the association between impairments in skeletal muscle microvascular oxygen delivery and cardiovascular blood flow regulation in ICU survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received mechanical ventilation for at least 7 days in the intensive care unit (ICU) and have subsequently been discharged from hospital.

Exclusion Criteria:

* Unable to provide consent
* Trajectory of health expected to be significantly limited in the upcoming 12 months
* those who self-report that they cannot climb at least one flight of stairs due to limited exercise capacity
* have significant orthopedic or musculoskeletal impairment affecting mobility
* have a medical history of neuromuscular disease
* ongoing respiratory limitations (i.e., supplemental oxygen)
* significant heart disease (i.e. ejection fraction less than 30%, unstable ischemic heart disease, severe valvular heart disease)
* a body mass index (BMI) of ≥ 40 kg/m2 (impacting NIRS signal due to adipose tissue thickness)
* if participant's primary residence is a significant distance from Winnipeg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU survivor: Patients who have received mechanical ventilation for at least 7 days in the intensive care unit (ICU) and have subsequently been discharged from hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
VO2 peak oxygen uptake | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  Peak Oxygen uptake (VO2, mL/kg/min) will be measured during incremental exercise on a cycle ergometer during cardiopulmonary exercise testing (CPET).
oxygen on/off kinetics | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  time constant (seconds) of oxygen uptake will be assessed at the transition to constant work rate exercise at the beginning of CPET; time constant (seconds) of oxygen uptake will also be assessed at the transition to rest at the end of CPET after reaching VO2 peak.
NIRS deoxygenation during exercise (deoxy-hemoglobin) | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  NIRS will be applied to the vastus lateralis during exercise testing. Deoxygenation profile, as measured by increase in deoxy-hemoglobin will be recorded throughout exercise. Higher values indicate impaired oxygen delivery to tissue.
NIRS deoxygenation during exercise (tissue saturation index) | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  NIRS will be applied to the vastus lateralis during exercise testing. Deoxygenation profile, as measured by decrease in tissue saturation index will be recorded throughout exercise. Lower values indicate impaired oxygen delivery to tissue.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) Questionnaire | Questionnaire will be conducted on up to 2 (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  will assess functional capacity, and will be administered by research staff. Response will be sought directly from the patient. FIM is scored with motor (13-91) and cognitive (5-35). Lower scores indicate lower functional independence
Frailty Index | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  The frailty index identifies 42 deficits, each coded as 0 (absent), 1 (present), or 0.5 (where intermediate values were possible). It was calculated as the cumulative proportion of deficits present (minimum score 0; maximum score 1.0), and then graded as mild (0 and 0.2), moderate (0.2 and 0.4) or severe frailty (>0.4). See references for studies where Index is derived.
Medical Research Council (MRC) sum score | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  Medical Research Council (MRC) sum score tests power in muscle groups for upper and lower extremities and score is tallied as the sum of all tested muscles. Value ranges from complete paralysis (0/60) to full strength (60/60). Score less than 48/60 denotes clinically significant weakness.
Anaerobic threshold | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  Work rate at anaerobic threshold (AT), represented at percentage of VO2 peak will be quantified with CPET. This corresponds to the time where oxygen (O2) utilization and carbon dioxide (CO2) production curves begin to diverge.
Forced Vital Capacity (FVC) | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  Standard spirometry techniques are used to quantify the maximum volume of expired breath (Litres), and represented as a %predicted compared to reference values. All tests are performed in accordance with standard ATS guidelines.
Forced Expiratory Volume at 1-second (FEV1) | Tests will be conducted on up to two (2) different occasions after ICU discharge: (i) 6 months, and (ii) 12 months.
  Standard spirometry techniques are used to quantify the volume of expired breath (Litres) in 1 second, and represented as a %predicted compared to reference values. All tests are performed in accordance with standard ATS guidelines.
Recruitment and retention | Ongoing throughout 12 months after ICU discharge
  The number of completed sessions within 12 months for each eligible patient will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Mendelson, MD PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Winnipeg, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendelson AA, Erickson D, Villar R. The role of the microcirculation and integrative cardiovascular physiology in the pathogenesis of ICU-acquired weakness. Front Physiol. 2023 May 10;14:1170429. doi: 10.3389/fphys.2023.1170429. eCollection 2023. PMID 37234410
- [Background] Heyland DK, Garland A, Bagshaw SM, Cook D, Rockwood K, Stelfox HT, Dodek P, Fowler RA, Turgeon AF, Burns K, Muscedere J, Kutsogiannis J, Albert M, Mehta S, Jiang X, Day AG. Recovery after critical illness in patients aged 80 years or older: a multi-center prospective observational cohort study. Intensive Care Med. 2015 Nov;41(11):1911-20. doi: 10.1007/s00134-015-4028-2. Epub 2015 Aug 26. PMID 26306719
- [Background] Muscedere J, Bagshaw SM, Boyd G, Sibley S, Norman P, Day A, Hunt M, Rolfson D. The frailty, outcomes, recovery and care steps of critically ill patients (FORECAST) study: pilot study results. Intensive Care Med Exp. 2022 Jun 10;10(1):23. doi: 10.1186/s40635-022-00446-7. PMID 35680740